CLINICAL TRIAL: NCT05585411
Title: PReventive Effect Of Left Bundle Branch Area Pacing Versus righT vEntricular paCing on All Cause deaTh, Heart Failure Progression, and Ventricular dysSYNChrony in Patients With Substantial Ventricular Pacing (PROTECT-SYNC): Multicenter Prospective Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2022-0824
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Bradyarrhythmia; Atrioventricular Block; Left Bundle Branch Area Pacing
Keywords: Left Bundle Branch Area pacing; Right Ventricular Pacing; Heart Failure; Atrioventricular block
MeSH Terms: conditions — Bradycardia; Atrioventricular Block; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBBAP group (Experimental): In this arm, a left bundle branch area pacing(LBBAP) lead will be attempted to be placed.
  Interventions: Procedure: Left bundle branch area pacing
- RVP group (Active Comparator): In this arm, a Right ventricular pacing (RVP) lead will be attempted to be placed.
  Interventions: Procedure: Right ventricular pacing

INTERVENTIONS:
Procedure: Left bundle branch area pacing — LBBAP success is defined if ventricular lead is successfully placed at interventricular septum and RBB configuration observed during unipolar tip pacing.
  LBB capture is defined if fulfilling criterion 1 and at least one in criteria 2.
  1. RBBB configuration observed during unipolar tip pacing
  2. One of the following should be met:
     1. Abrupt shortening of Stim-LVAT (stimulus to peak of the R wave in V6 [LV activation time]) of >10ms during increasing output
     2. Short and constant stim-LVAT and the shortest stim-LVAT <75ms in non-LBBB and <85ms in LBBB
     3. Programmed stimulation by pacing lead changes QRS morphology from nonselective LBB to LV septal capture
     4. LBB potential (LBB-V interval of 15 to 35ms)
     5. Transition from nonselective LBB capture to selective LBB capture at near threshold outputs
  If criterion 1 is fulfilled but none in criteria 2 is met, the procedure is considered to be deep septal pacing (DSP).
  Arms: LBBAP group
Procedure: Right ventricular pacing — Right ventricular pacing is the traditional pacing modality for ventricular pacing. Implantation of a RV pacing lead (apex or septum of right ventricle) will be attempted using the standard-of-care technique first
  Arms: RVP group

SUMMARY:
PROTECT-SYNC study is a multicenter, randomized, controlled trial. A total of 7 medical centers across Republic of Korea will enroll 450 patients during 2 years of enrollment period, and followed for 2 years of follow-up period. The purpose of this study to compare the clinical outcomes of Left Bundle Branch Area Pacing (LBBAP) compared to Right Ventricular Pacing (RVP) in bradyarrhythmia patients who require high burden of ventricular pacing (>40%).

DETAILED DESCRIPTION:
PROTECT-SYNC study is a multicenter, randomized, controlled trial that is designed to assess whether LBBAP may reduce the risk of composite primary endpoint including all cause mortalty, HF hospitalization and/or urgent HF related visit, occurrence of pacing induced CMP, and CRT-upgrade event, compared to RVP in patients who require substantial (>40%) ventricular pacing. Patients who require pacemaker and substantial (>40%) ventricular pacing will be randomized to LBBAP or RVP group, and a total of 7 medical centers across Republic of Korea will enroll 450 patients during 2 years of enrollment period, and followed for 2 years of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years old and willing and capable to give informed consent
2. Patients who is willing and able to comply with the prescribed follow-up tests and schedule of evaluations.

3 Scheduled to receive a pacemaker implant 4. Substantial percentage of V pacing rate (>40%) is anticipated

Exclusion criteria:

1. Incapacitated or unable to read or write
2. Patient who is an indication of ICD or CRT
3. History of prosthetic valve surgery on tricuspid valve
4. Prior myocardial infarction including ventricular septum
5. Life expectancy < 12 months due to any condition
6. Unavailable for at least 24 months of follow-up visits
7. Pregnant or breastfeeding at the time of signing consent
8. Prior Heart transplant surgery
9. Persistent Left Superior Vena Cava (PLSVC)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
composite of all-cause death, heart failure hospitalization, occurrence of pacing induced cardiomyopathy, and an upgrade to cardiac resynchronization therapy | during 2 years after pacemaker implantation
  All-cause death: including cardiovascular and non-cardiovascular deaths.
  Heart failure hospitalization: An unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required intravenous therapy.
  Occurrence of Pacing induced cardiomyopathy : LVEF <50% and absolute LVEF decline ≥10% or increase in LVESV ≥15% Upgrade to cardiac resynchronization therapy (CRT): Upgrade from pacemaker to CRT-Pacemaker/CRT-Defibrillator due to impaired LV function (LVEF decrease to 40% or less).

SECONDARY OUTCOMES:
all cause mortality | during 2 years after pacemaker implantation
  All cause deaths including cardiovascular and non-cardiovascular deaths.
Cardiovascular mortality | during 2 years after pacemaker implantation
  Cardiovascular death
Heart failure hospitalization | during 2 years after pacemaker implantation
  An unplanned outpatient or emergency department visit or inpatient hospitalization in which the patient presented with signs and symptoms consistent with heart failure and required intravenous therapy.
success rate of LBBAP implantation | during 3days after pacemaker implantation
  LBBAP success is defined if ventricular lead is successfully placed at interventricular septum and RBB configuration observed during unipolar tip pacing.
LBBAP related complications | during 2 years after pacemaker implantation
  Loss of lead function or need for lead revision, extraction, replacement for any reason
LBB capture failure | during 2 years after pacemaker implantation
  failed LBB capture, confirmed by investigator
Short-term procedure and Device related complications | during 1wk after pacemaker implantation
  composite of device and procedure related complications until 7 days after procedure
Long-term procedure and Device related complications | during 1wk after pacemaker implantation
  composite of device and procedure related complications after 7 days after procedure
Rate of LV systolic dysfunction | 6month and 2yr after pacemaker implantation
  LVEF <50% and absolute reduction in LVEF >10%, and/or an increase in LVESV ≥15%.
Changes in cardiopulmonary exercise test parameters | 6month and 2yr after pacemaker implantation
  (VO2 peak, Exercise intensity, Peak Respiratory Exchange Ratio (Peak RER), Exercise time, age predicted aerobic capacity, VE/VCO2 slope, Lactate threshold, Max predicted HR, Max HR / Max predicted HR, presence of ST change , AF at Baseline, Incident AF during exercise
Incidental atrial fibrillation | during 2 years after pacemaker implantation
  Newly developed atrial fibrillation in patients without documented atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: TaeHoon Kim, Principal Investigator — Severance Cardiovascular Hospital Yonsei University
Locations (8):
- South Korea (8):
  - Bucheon Sejong Hospital, Bucheon-si
  - GyeongSang National University Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Chungju
  - Asan Medical Center, Seoul
  - Kyunghee University hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tops LF, Schalij MJ, Bax JJ. The effects of right ventricular apical pacing on ventricular function and dyssynchrony implications for therapy. J Am Coll Cardiol. 2009 Aug 25;54(9):764-76. doi: 10.1016/j.jacc.2009.06.006. PMID 19695453
- [Background] Tse HF, Lau CP. Long-term effect of right ventricular pacing on myocardial perfusion and function. J Am Coll Cardiol. 1997 Mar 15;29(4):744-9. doi: 10.1016/s0735-1097(96)00586-4. PMID 9091519
- [Background] Sweeney MO, Hellkamp AS, Ellenbogen KA, Greenspon AJ, Freedman RA, Lee KL, Lamas GA; MOde Selection Trial Investigators. Adverse effect of ventricular pacing on heart failure and atrial fibrillation among patients with normal baseline QRS duration in a clinical trial of pacemaker therapy for sinus node dysfunction. Circulation. 2003 Jun 17;107(23):2932-7. doi: 10.1161/01.CIR.0000072769.17295.B1. Epub 2003 Jun 2. PMID 12782566
- [Background] Wilkoff BL, Cook JR, Epstein AE, Greene HL, Hallstrom AP, Hsia H, Kutalek SP, Sharma A; Dual Chamber and VVI Implantable Defibrillator Trial Investigators. Dual-chamber pacing or ventricular backup pacing in patients with an implantable defibrillator: the Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial. JAMA. 2002 Dec 25;288(24):3115-23. doi: 10.1001/jama.288.24.3115. PMID 12495391
- [Background] Abdelrahman M, Subzposh FA, Beer D, Durr B, Naperkowski A, Sun H, Oren JW, Dandamudi G, Vijayaraman P. Clinical Outcomes of His Bundle Pacing Compared to Right Ventricular Pacing. J Am Coll Cardiol. 2018 May 22;71(20):2319-2330. doi: 10.1016/j.jacc.2018.02.048. Epub 2018 Mar 10. PMID 29535066
- [Background] Kusumoto FM, Schoenfeld MH, Barrett C, Edgerton JR, Ellenbogen KA, Gold MR, Goldschlager NF, Hamilton RM, Joglar JA, Kim RJ, Lee R, Marine JE, McLeod CJ, Oken KR, Patton KK, Pellegrini CN, Selzman KA, Thompson A, Varosy PD. 2018 ACC/AHA/HRS Guideline on the Evaluation and Management of Patients With Bradycardia and Cardiac Conduction Delay: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Circulation. 2019 Aug 20;140(8):e382-e482. doi: 10.1161/CIR.0000000000000628. Epub 2018 Nov 6. No abstract available. PMID 30586772
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Mao G, Vijayaraman P, Ellenbogen KA. Long-term outcomes of His bundle pacing in patients with heart failure with left bundle branch block. Heart. 2019 Jan;105(2):137-143. doi: 10.1136/heartjnl-2018-313415. Epub 2018 Aug 9. PMID 30093543
- [Background] Vijayaraman P, Ponnusamy S, Cano O, Sharma PS, Naperkowski A, Subsposh FA, Moskal P, Bednarek A, Dal Forno AR, Young W, Nanda S, Beer D, Herweg B, Jastrzebski M. Left Bundle Branch Area Pacing for Cardiac Resynchronization Therapy: Results From the International LBBAP Collaborative Study Group. JACC Clin Electrophysiol. 2021 Feb;7(2):135-147. doi: 10.1016/j.jacep.2020.08.015. Epub 2020 Oct 28. PMID 33602393
- [Background] Sharma PS, Patel NR, Ravi V, Zalavadia DV, Dommaraju S, Garg V, Larsen TR, Naperkowski AM, Wasserlauf J, Krishnan K, Young W, Pokharel P, Oren JW, Storm RH, Trohman RG, Huang HD, Subzposh FA, Vijayaraman P. Clinical outcomes of left bundle branch area pacing compared to right ventricular pacing: Results from the Geisinger-Rush Conduction System Pacing Registry. Heart Rhythm. 2022 Jan;19(1):3-11. doi: 10.1016/j.hrthm.2021.08.033. Epub 2021 Sep 3. PMID 34481985
- [Background] Curtis AB, Worley SJ, Adamson PB, Chung ES, Niazi I, Sherfesee L, Shinn T, Sutton MS; Biventricular versus Right Ventricular Pacing in Heart Failure Patients with Atrioventricular Block (BLOCK HF) Trial Investigators. Biventricular pacing for atrioventricular block and systolic dysfunction. N Engl J Med. 2013 Apr 25;368(17):1585-93. doi: 10.1056/NEJMoa1210356. PMID 23614585